CLINICAL TRIAL: NCT03820206
Title: The Value of Tranxemic Acid to Reduce Intraoperative Blood Loss During Elective Cesarean Sections in High Risk Women: A Randomized Controlled Trial
Brief Title: The Value of Tranxemic Acid to Reduce Intraoperative Blood Loss During Elective Cesarean Sections in High Risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 50
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid group (Active Comparator): 1 g (10 mL) tranexamic acid (Kapron, Amoun, Egypt; stored in a dry container at 15 °C-30 °C) diluted in 20 mL of 5% glucose slowly administered intravenously 15 minutes before skin incision over a 5-minute period.
  Interventions: Drug: Tranexamic Acid; Procedure: Cesarean section
- Control group (Placebo Comparator): 30 mL of 5% glucose slowly administered intravenously 15 minutes before skin incision over a 5-minute period.
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Drug: Tranexamic Acid — 1 g (10 mL) tranexamic acid stored in a dry container at 15 °C-30 °C) diluted in 20 mL of 5% glucose slowly administered intravenously 15 minutes before skin incision over a 5-minute period.
  Other Names: Kapron
  Arms: Tranexamic acid group
Procedure: Cesarean section — Lower segement transverse cesarean section
  Other Names: Lower segment elective cesarean section

SUMMARY:
A full medical history will be obtained from all participants. Obstetric ultrasonography and laboratory tests will be performed.According to group assignment, either 1 g(10 mL) tranexamic acid stored in a dry container at 15 °C-30 °C) diluted in 20 mL of 5% glucose or 30 mL of 5% glucose will be slowly administered intravenously 15 minutes before skin incision over a 5-minute period.

Following delivery, patients in both groups will receive an intravenous bolus of 5 IU oxytocin , 1 mL(0.2 mg) intramuscular ergometrine , and 20 IU oxytocin in 500 mL lactated Ringer's solution(infused at a rate of 125 mL/h)

DETAILED DESCRIPTION:
A full medical history will be obtained from all participants. Obstetric ultrasonography and laboratory tests will be performed, including prothrombin time, prothrombin concentration, complete blood count, and liver and kidney function tests. Maternal body weight and vital signs (heart rate, blood pressure, and respiratory rate) will be checked 30 minutes before surgery. According to group assignment, either 1 g(10 mL) tranexamic acid (Kapron, Amoun, Egypt; stored in a dry container at 15 °C-30 °C) diluted in 20 mL of 5% glucose or 30 mL of 5% glucose will be slowly administered intravenously 15 minutes before skin incision over a 5-minute period.

Following delivery, patients in both groups will receive an intravenous bolus of 5 IU oxytocin (Syntocinon, Novartis, Basel, Switzerland), 1 mL(0.2 mg) intramuscular ergometrine (Methergin, Novartis, Basel, Switzerland), and 20 IU oxytocin in 500 mL lactated Ringer's solution(infused at a rate of 125 mL/h).

Fluid monitoring will be performed through rate of infusion and urine output. A complete blood count test will be performed 24 hours after delivery. On discharge, patients who received tranexamic acid will be given a brief orientation regarding symptoms and signs of a thromboembolic event and will be instructed to contact the investigators immediately if any occurred.

All patients will be examined for thromboembolic events at the 1- and 4-week follow-up visits

EBL will be calculated according to the formula:

EBL = EBV x Preoperative hematocrit-Postoperative hematocrit Preoperative hematocrit where EBV is estimated blood volume (mL; weight in kg × 85). For a two-tailed test at an α level of 0.05, the difference between the two groups regarding the primary outcome measure (EBL) had a power of 1.0 (100%) in a post hoc calculation.

ELIGIBILITY:
Inclusion Criteria:

* • Grand multipara

  * Multiple pregnancy
  * Polyhydraminos (AFI is more than 24 cm).
  * Placenta previa
  * Gestational diabetes mellitus
  * Preeclampsia
  * Anemia complicating pregnancy (Hemoglobin is less than 11 gm/dl)

Exclusion Criteria:

* • Allergy to tranxemic acid.

  * H/o suggestive of bleeding disorders
  * previous history of deep vein thrombosis
  * Abnormally invasive placenta
  * Emergency cesarean sections
  * Intraoprative complications during cesarean sections as uterine artery injury and broad ligamentary hematoma.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss (EBL) during cesarean delivery | during the operation
  EBL will be calculated according to the formula:
  EBL = EBV x Preoperative hematocrit-Postoperative hematocrit Preoperative hematocrit where EBV is estimated blood volume (mL; weight in kg × 85)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shalaby MA, Maged AM, Al-Asmar A, El Mahy M, Al-Mohamady M, Rund NMA. Safety and efficacy of preoperative tranexamic acid in reducing intraoperative and postoperative blood loss in high-risk women undergoing cesarean delivery: a randomized controlled trial. BMC Pregnancy Childbirth. 2022 Mar 14;22(1):201. doi: 10.1186/s12884-022-04530-4. PMID 35287618